## NUTRITIONAL STATUS ASSESSMENT OF PEDIATRIC CYSTIC FIBROSIS PATIENTS AND EFFECT OF NUTRITION EDUCATION ON NUTRITIONAL STATUS

STUDY PROTOCOL DATE: 03.09.2021

| Follow-<br>up | EDUCATION GROUP | CONTROL GROUP |
|---|---|---|
| Meet | <ul> <li>Introduction, explanation of the purpose of the research, giving information about the practices and obtaining informed consent</li> <li>Application of questionnaires and scales</li> <li>Education for the family: How to keep a correct and proper record of food consumption? (Using Food &amp; Food Photo Catalog)</li> </ul> | <ul> <li>Introduction, explanation of the purpose of the research, giving information about the practices and obtaining informed consent</li> <li>Application of questionnaires and scales</li> <li>Education for the family: How to keep a correct and proper record of food consumption? (Using Food &amp; Food Photo Catalog)</li> </ul> |
| 1st<br>Week | Cystic Fibrosis Nutrition Education-I: The<br>Importance of Healthy Nutrition, Carbohydrate,<br>Fat, Protein, Vitamin-Minerals, Water. | |
| | <ul> <li>Definition of healthy eating,</li> </ul> | |
| | The importance of adequate energy and | |
| | macro-micronutrient intake for CF patients, | |
| | <ul> <li>Foods containing macro and micronutrients</li> </ul> | |
| | such as carbohydrate-fat-protein-vitamin-mineral | |
| 2nd | Cystic Fibrosis Nutrition Education-II: Food | |
| Week | Groups, Common Nutritional Problems by Age | |
| | Groups and Solution Suggestions. | |
| | The four basic food groups and the nutrients they | |
| | <ul><li>contain</li><li>Changelists in TÜBER</li></ul> | |
| | <ul> <li>Changensis in TOBER</li> <li>Common nutritional problems according to age</li> </ul> | |
| | groups and solution suggestions | |
| 3rd | | |
| Week | Cystic Fibrosis Nutrition Education-III: General Review and Frequently Asked Questions and Answers | |
| | <ul> <li>Summary information about the first two trainings,</li> <li>Recommendations on how children diagnosed with</li> </ul> | |
| | CF can increase their energy and fat intake | |
| | • Things to consider about PERT treatment | |
| | Frequently asked questions and answers | |
| | Document sharing | |
| 1st | <ul> <li>Application of questionnaires and scales</li> </ul> | <ul> <li>Application of questionnaires and</li> </ul> |
| month | <ul> <li>Collection of food records</li> </ul> | scales |
| and 3rd<br>month | | <ul> <li>Collection of food records</li> </ul> |